CLINICAL TRIAL: NCT00961194
Title: Evaluation of the Analgesic Effect of Orally Administrated Ketamine in Peripheral Neuropathic Pain Disease: Comparison of Three Doses Versus Placebo.
Brief Title: Oral Ketamine Administration in Patients With Peripheral Neuropathic Pain
Acronym: KETACLUD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 0730102; AOL 2007 (Other: AOL 2007)
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Neuropathic Pain
Keywords: Ketamine; pain; neuropathic pain; chronic
MeSH Terms: conditions — Neuralgia; Pain; Bronchiolitis Obliterans Syndrome | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator): The study will be conducted using 4 parallel groups (three doses of ketamine versus placebo).Each patient will receive the indicated dose of oral ketamine or placebo once and if there are not adverse events, he will be able to continue the treatment three times a day, during 7 days (between visit 2 and 3).
  The oral ketamine will be administered in form of syrup.
  Interventions: Drug: Ketamine
- dose of ketamine tested = 0.35 mg/kg (Experimental): The study will be conducted using 4 parallel groups (three doses of ketamine versus placebo).Each patient will receive the indicated dose of oral ketamine or placebo once and if there are not adverse events, he will be able to continue the treatment three times a day, during 7 days (between visit 2 and 3).
  The oral ketamine will be administered in form of syrup.
  Interventions: Drug: Ketamine
- dose of ketamine tested = 0.7 mg/kg (Active Comparator): The study will be conducted using 4 parallel groups (three doses of ketamine versus placebo).Each patient will receive the indicated dose of oral ketamine or placebo once and if there are not adverse events, he will be able to continue the treatment three times a day, during 7 days (between visit 2 and 3).
  The oral ketamine will be administered in form of syrup.
  Interventions: Drug: Ketamine
- dose of ketamine tested = 1.4 mg/kg (Active Comparator): The study will be conducted using 4 parallel groups (three doses of ketamine versus placebo).Each patient will receive the indicated dose of oral ketamine or placebo once and if there are not adverse events, he will be able to continue the treatment three times a day, during 7 days (between visit 2 and 3).
  The oral ketamine will be administered in form of syrup.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Initial dosage: 250 mg/5 ml
  Three doses of ketamine will be tested:
  * 0.35 mg/kg
  * 0.7 mg/kg
  * 1.4 mg/kg Each patient will receive the indicated dose of oral ketamine or placebo once and if there are not adverse events, he will be able to continue the treatment three times a day, during 7 days (between visit 2 and 3).
  The oral ketamine will be administered in form of syrup.
  Other Names: Ketamine PANPHARMA

SUMMARY:
Nowadays, available drugs cannot always produce pain relief in patients with neuropathic pain disease.

It is believed that drugs acting as antagonists of the N-methyl-D-aspartic acid (NMDA) receptor may have been efficient in the treatment of neuropathic pain disorders.

Ketamine is the only NMDA receptor antagonist commercially available in France. Ketamine is usually administered intravenously for surgical anesthesia.

The intravenous administration of ketamine will be difficult to manage in the treatment of chronic neuropathic pain.

Some trials using oral ketamine for the treatment of neuropathic pain were conducted but results were heterogeneous. This may be explained by the different range of ketamine doses tested.

The aim of this clinical trial is to identify a safe and an efficient dose of orally administrated ketamine for the treatment of peripheral neuropathic pain.

The clinical trial will be conducted in Toulouse Hospital, France. This study is a randomized, double-blind, placebo-controlled trial. The study will be conducted using 4 parallel groups (three doses of ketamine versus placebo).

DETAILED DESCRIPTION:
In previous studies, it was shown that when ketamine was administrated by the intravenous route, its analgesic action was rapid. In one study, when oral ketamine was administrated to patients suffering from neuropathic pain, in six out of nine patients, pain was relieved after 24 hours post-administration.

In this study, ketamine will be administrated during seven days, which will allow us to evaluate ketamine efficiency and safety.

The effect of ketamine on pain intensity will be mainly studied using a visual analogue scale (VAS) but also taking into account the score assigned by the patient to his pain. This score will be noted down by patients before, during and after ketamine treatment.

Evaluation of benefit/risk for ketamine administration during this trial, shows that even if adverse events are not excluded, the benefit for the patients may be neuropathic pain relief.

Because clinical current knowledge regarding oral administration of ketamine is limited, this trial intends to enlarge information about ketamine efficiency and safety, more particularly in neuropathic pain disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients must suffer from peripheral neuropathic chronic pain.
* Pain score must be at least 40 mm in a VAS (reflecting pain intensity during the 7 days and the day before visit 1).
* Patients in which pain is not satisfactory relieved by level 1, 2 or 3 analgesic drugs (associated or not with antidepressants or antiepileptic drugs). Patients treated with level 2 or 3 analgesic drugs must stop these treatments one week before and during ketamine treatment.
* Patients must benefit from the French Social security system.
* Patients must be able to complete the tests.
* Patients must give a written informed consent.
* Patients must be aged from 30 to 90 years.
* Female fertile patients must use an efficient method of contraception.

Exclusion Criteria:

* Patients not suffering from peripheral neuropathic chronic pain.
* Pain score is less than 40 mm in a VAS (reflecting pain intensity during the 7 days and the day before visit 1).
* Patients not able to complete the tests.
* Patients not able to stop level 2 or 3 analgesic drugs.
* Patients in which ketamine is contraindicated:

  * Hypersensibility to one of the compounds of the ketamine syrup
  * Uncontrolled arterial hypertension
  * Recent cardio vascular accident
  * Severe cardiac problems
  * Drug abuse
  * Psychosis

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-03; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain intensity using a 10 cm visual analogue scale (VAS) (0 = no pain; 10 = worst possible pain) before and after 7 days of oral administration of one of the three doses of ketamine or placebo. | V1 (14 days before ketamine treatment), at V2 (before oral administration of one of the three doses of ketamine or placebo), at V3 (after 7 days of oral administration), and at V4 (after 7 days of the end of treatment)

SECONDARY OUTCOMES:
Pain intensity will be evaluated by measuring thermal sensibility. A thermode will be used to determine the heat and cold pain thresholds (thermotest) and by measuring hyperalgesia | Thermotest and hyperalgesia will be assessed at T0 and T1 hour, at visit 2 and visit 3

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Cantagrel, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Service de Neurochirurgie, Toulouse, France